CLINICAL TRIAL: NCT01351311
Title: Assessment of Effectiveness of Resistance Training Exercise Using the Swiss Ball in Patients With Ankylosing Spondylitis
Brief Title: Resistance Training Exercise Using the Swiss Ball in Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, MsC, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDAAAMC
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Ankylosing Spondylitis
Keywords: treatment; exercise; resistance training; swiss ball; functional capacity
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity | interventions — Exercise; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Group (Experimental): Resistance exercise with swiss ball and drug treatment
  Interventions: Other: Exercise
- Control Group (Other): Drug treatment
  Interventions: Other: Drug treatment

INTERVENTIONS:
Other: Exercise — Resistance Training exercise with swiss ball
  Other Names: Experimental group
  Arms: Exercise Group
Other: Drug treatment — Drug treatment
  Other Names: Control group
  Arms: Control Group

SUMMARY:
The aim of the present study is to assess the effectiveness of resistance training with swiss ball in the treatment of patients with ankylosing spondylitis.

DETAILED DESCRIPTION:
A randomized, controlled, single-blind, prospective trial being conducted involving 54 patients with ankylosing spondylitis, selected from outpatient clinics - UNIFESP. They will be randomized in intervention group (n = 27) conduct training for muscle strengthening with the aid of the Swiss ball and in the control group (n = 27) did not undergo any intervention. Eight exercises will be conducted with intent to engage all muscle groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of AS steinbrocker functional class I-II
* Basic medication stable for at least three months
* Agreed to participate and signed term of informed consent

Exclusion Criteria:

* Uncontrolled hypertension
* Coronary artery disease
* History of revascularization
* History of syncope or arrhythmias induced by exercise
* Decompensated diabetes mellitus
* Severe psychiatric illness
* Fibromyalgia
* Another medical condition more disabling than AS
* History of exercise regular (at least 30 minutes 2 times per week)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Functional Index (BASFI) | 16 weeks
  Functional capacity assessed by BASFI

SECONDARY OUTCOMES:
LIKERT SCALE | 16 weeks
  Likert scale by patients.
1 REPETITION MAXIMUM TEST | 16 weeks
  muscle strength by testing an repetition maximum (1 RM)
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 16 weeks
  disease activity by BASDAI (The Bath Ankylosing Spondylitis Disease Activity Index)
Bath Ankylosing Spondylitis Metrology Index (BASMI) | 16 weeks
  spinal mobility by BASMI
erythrocyte sedimentation rate (ESR) | 16 weeks
6-MINUTE WALK TEST | 16 weeks
TIME UP AND GO TEST | 16 weeks
Short form-36 (SF-36) | 16 weeks
  quality of life by SF-36
QUANTITY OF ANALGESICS AND ANTI-INFLAMATORY USED | 16 weeks
Health Assessment Questionnaire (HAQ) Health Assessment Questionnaire | 16 weeks
  Function

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Souza, PT, MSc, Principal Investigator — Federal University of São Paulo; Fábio Jennings, MD, MSc, Study Director — Federal University of São Paulo; Jamil Natour, MD, PHD, Study Chair — Division of Rheumatology, Federal University of Sao Paulo
Locations (1):
- Marcelo Cardoso de Souza, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Derived] Souza MC, Jennings F, Morimoto H, Natour J. Swiss ball exercises improve muscle strength and walking performance in ankylosing spondylitis: a randomized controlled trial. Rev Bras Reumatol Engl Ed. 2017 Jan-Feb;57(1):45-55. doi: 10.1016/j.rbre.2016.09.009. Epub 2016 Oct 20. English, Portuguese. PMID 28137402